CLINICAL TRIAL: NCT04627168
Title: The Effects of Transcutaneous Abdominal Stimulation on Bowel Function in Persons With Spinal Cord Injury and in Able-bodied Persons With Chronic Constipation.
Brief Title: Trancutaneous Abdominal Stimulation on Bowel Function.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amol Soin, M.D., MBA (Other)
Responsible Party: Sponsor-Investigator, Amol Soin, M.D., MBA, Medical Director, Ohio Pain Clinic
Organization: Ohio Pain Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM 100-1
Record Dates: First submitted 2020-11-01; First posted 2020-11-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injuries; Constipation
Keywords: spinal cord injury; stimulation; constipation
MeSH Terms: conditions — Spinal Cord Injuries; Constipation

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to 1 of 2 groups. The first subject group will include spinal cord injured persons presenting with constipation, the second group - able-bodied persons with chronic constipation. In both groups, subjects will receive transcutaneous abdominal electrical stimulation that will be delivered through commercially available equipment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Spinal cord injured persons (Experimental): Persons living with spinal cord injury presenting with constipation due to neurogenic bowel dysfunction.
  Interventions: Device: Non-invasive, surface electrical stimulation device, DS5 Digitimer
- Persons without neurogenic bowel dysfunction (Experimental): Abled-bodied persons with chronic constipation.
  Interventions: Device: Non-invasive, surface electrical stimulation device, DS5 Digitimer

INTERVENTIONS:
Device: Non-invasive, surface electrical stimulation device, DS5 Digitimer — Transcutaneous abdominal electrical stimulation will be delivered through the commercially available equipment, a DS5 Digitimer.

SUMMARY:
This is a prospective, single-center, feasibility study to determine the sensations elicited by non-invasive abdominal electrical stimulation and its effects on bowel function in spinal cord injured individuals and in able-bodied persons with chronic constipation. Electrical stimulation will be delivered through commercially available equipment to each subject during a single site visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, treatment feasibility study to determine the efficacy of electrical stimulation for bowel functions. The study will determine sensations elicited by non-invasive, transcutaneous abdominal electrical stimulation and its effects on bowel function in spinal cord injured individuals and in able-bodied persons with chronic constipation. The electrical stimulation will be delivered through commercially available equipment to each subject during a single site visit. Visits are anticipated to be no more than 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* For spinal cord injury subject group:

  * Traumatic or non-traumatic spinal cord injury;
  * Constipation;
  * Motor-complete or motor-incomplete spinal cord injury;
  * Quadriplegia or paraplegia;
  * Post-injury time ≥ 1 year;
  * Neurogenic Bowel Dysfunction Score ≥ 7.
* For able-bodied subject group:

  * Diagnosis of intestinal constipation according to the Rome IV criteria;
  * Chronic constipation as defined by < 3 bowel movements per week for > 3 months.
* For both subject groups:

Can read, understand and willingly sign an Institutional Review Board approved informed consent document that describes the study's risks and benefits.

Exclusion Criteria:

1. Presence of any organic cause for intestinal constipation;
2. Have chronic fecal incontinence;
3. Have skin infection/lesion in the area of electrode application or systemic skin disease;
4. Have an implanted electronic device (such as heart pacemaker, insulin or baclofen pump, etc);
5. Have symptomatic cardiac disease;
6. Have uncontrolled diabetes;
7. Presence of abdominal hernia;
8. Have a stoma, rectal tear, or untreated hemorrhoids;
9. Have a significant psychiatric disorder;
10. For female subjects, being pregnant, actively planning a pregnancy or breast-feeding a child;
11. Be participating in another clinical study that would confound data analysis;
12. Have a cognitive impairment or exhibits any characteristic that would limit the study candidate's ability to complete study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Duration of the occurrence of first stool | 7 days
  The time between the onset of transcutaneous abdominal electrical stimulation and the first stool will be measured.
Total defecation time (duration) | 7 days
  The time (duration) to complete total defecation following the stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Soin, MD, Principal Investigator — Ohio Pain Clinic
Locations (1):
- Ohio Pain Clinic, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No